CLINICAL TRIAL: NCT02045472
Title: Double-Blind, Placebo-Controlled, Dose-Escalation Phase 1 Study in Healthy Volunteers to Evaluate the Safety and Pharmacokinetics of a Human Monoclonal Antibody (VIS410) to Influenza Type A Hemagglutinin
Brief Title: A Study of VIS410 to Assess Safety and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIS-C001
Record Dates: First submitted 2014-01-21; First posted 2014-01-24 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Influenza
Keywords: Influenza; Monoclonal antibody
MeSH Terms: conditions — Influenza, Human | interventions — VIS410 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIS410 (Experimental): VIS410 administered as a single infusion with ascending dose-escalation ranging from 2 to 50 mg/kg
  Interventions: Drug: VIS410
- Placebo (Placebo Comparator): Placebo administered as a single infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIS410
  Arms: VIS410
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, immunogenicity and pharmacokinetics of single escalating doses of VIS410 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Body mass index between 18 and 33 kg/m2, inclusive
* Normal labs
* Volunteers agree to use acceptable contraceptive measures

Exclusion Criteria:

* Prior receipt of antibody or biologic therapy
* History of cancer, heart disease, diabetes, respiratory condition (eg asthma), autoimmune disorder, blood dyscrasias
* Any chronic condition requiring daily prescription or over the counter medication
* History of a previous severe allergic reaction
* Drug or alcohol abuse within previous 12 months
* Positive serology for human immunodeficiency virus (HIV) antibody, hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg)
* Positive pregnancy test
* Breast feeding
* Positive drug or alcohol test at screening or check-in
* Receipt of licensed vaccine (within 30 days) or other investigational product within 30 days or 5 half-lives, whichever is longer, before study product administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety assessment | 120 days post-infusion
  Incidence of adverse events

SECONDARY OUTCOMES:
Pharmacokinetic analysis | 56 days post-infusion
  Serum concentration-time profile
Immunogenicity | 120 days post-infusion
  Detect and measure anti-drug antibodies to VIS410

CONTACTS AND LOCATIONS:
Overall Officials: J K Berg, MD, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Wollacott AM, Boni MF, Szretter KJ, Sloan SE, Yousofshahi M, Viswanathan K, Bedard S, Hay CA, Smith PF, Shriver Z, Trevejo JM. Safety and Upper Respiratory Pharmacokinetics of the Hemagglutinin Stalk-Binding Antibody VIS410 Support Treatment and Prophylaxis Based on Population Modeling of Seasonal Influenza A Outbreaks. EBioMedicine. 2016 Feb 26;5:147-55. doi: 10.1016/j.ebiom.2016.02.021. eCollection 2016 Mar. PMID 27077121